CLINICAL TRIAL: NCT05451147
Title: A Comparative Study of the Effect of "Chhinnavahni Kashaya Vati" Along With "Agnimantha Kwatha" & Metformin in the Management of Madhumeha w.s.r. to Diabetes Mellitus (Type II)
Brief Title: A Comparative Study of the Effect of Ayurvedic Drugs and Metformin in the Management of Diabetes Mellitus (Type II)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: A & U Tibbia College Karol Bagh (Other)
Responsible Party: Principal Investigator, Dr. Richa Bhardwaj, PG Scholar (Kayachikitsa), A & U Tibbia College Karol Bagh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N.F.5(283)/2013-CO
Record Dates: First submitted 2022-05-29; First posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Randomized, Controlled, Parallel Group Trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): DRUG: Chhinnavahni Kashaya Vati FORM: Tablet DOSE: 1 g TDS (2 Tab. of 500 mg each), Before Meals MODE OF ADMINISTRATION: Oral ANUPAAN: 20 ml of Agnimantha Kwatha DURATION: 3 Months
  Interventions: Drug: Chhinnavahni Kashaya Vati along with Agnimantha Kwatha
- GROUP B (Active Comparator): DRUG: Metformin FORM: Tablet DOSE: 500mg BID/TDS, Before Meals MODE OF ADMINISTRATION: Oral ANUPAAN:: Plain Water DURATION 3 Months
  Interventions: Drug: Metformin Hydrochloride

INTERVENTIONS:
Drug: Chhinnavahni Kashaya Vati along with Agnimantha Kwatha — Drug: Chhinnavahni Kashaya Vati Form : Tablet Dose: 1g TDS (2x500 mg), Before meals Mode of Administration: Oral Anupaan: 20 ml of Agnimantha Kwatha Duration: 3 Months
  Other Names: Chhinnavahni Kashaya Vati; Agnimantha Kwatha
  Arms: Group A
Drug: Metformin Hydrochloride — Drug: Metformin Form: Tablet Dose: 500mg BID/TDS, Before meals Mode of Administration: Oral Anupaan: Plain water Duration: 3 Months
  Other Names: Metformin
  Arms: GROUP B

SUMMARY:
Present study entitled "A Comparative Study of the Effect of "Chhinnavahni Kashaya Vati" along with "Agnimantha Kwatha" & Metformin in the management of Madhumeha w.s.r. to Diabetes mellitus (Type II)" is a small effort to find out an effective remedy for Madhumeha i.e. Diabetes Mellitus Type-2

DETAILED DESCRIPTION:
Single centered, randomized clinical trial of Chhinnavahni Kashaya Vati along with Agnimantha Kwatha was carried out on total of 60 registered patients. They were randomly classified in two groups, where in Group-A received Chhinnavahni Kashaya Vati with Agnimantha Kwatha and Group-B received Metformin for 12 weeks. Out of these, 12 patients did not complete the full course of the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either sex aged between 20 to 60 years.
2. If yes in any two of the four:

   * Blood sugar -fasting > 126 and ≤ 250 mg/dl.
   * PP > 200 mg/dl and ≤350 mg/dl.
   * Glycosylated Haemoglobin (HbA1c) > 6.5% and < 9%.
   * Subjects having classical symptoms of diabetes with random glucose levels ≥200mg/dl (≤350mg/dl).
3. Diagnosed cases of Type II Diabetics having Glycosylated Haemoglobin (HbA1c) between 6.5-9% without or {with metformin in a dose1g-1.5g/day (for Group-B)}.
4. Subjects who are able to come for follow up on fixed visits and are well aware about the treatment plan.
5. Subjects willing to participate and able to provide written informed consent.

Exclusion Criteria:

1. Age below 20 and above 60yrs.
2. Subject of Type-I DM (insulin dependent DM) or Type-II DM on insulin/OHA's other than metformin/ any other AYUSH medication for glucose control.
3. Subjects suffering from the complications of Diabetes mellitus viz., diabetic neuropathy, diabetic nephropathy, diabetic retinopathy etc. which require an urgent treatment.
4. Uncontrolled Hypertensive subjects (BP with or without medication >140/90 mmHg after 5 mins of rest).
5. Subjects with any unstable Heart disease or known cases of MI, unstable angina or CHF.
6. Patients with concurrent Hepatic Dysfunction (defined as AST and/or ALT > 2 times of the upper normal limit) or Renal Dysfunction, uncontrolled Pulmonary Dysfunction (asthmatic and COPD subjects).
7. Subjects with current or past diagnosis of malignancy (any malignancy diagnosis in last five years).
8. Subjects who have a recent history or who are currently known to abuse of alcohol or drugs.
9. Subjects suffering from major systemic illness necessitating long term drug treatment (Rheumatoid arthritis, Psycho-Neuro-Endocrinal disorders, TB, AIDS etc).
10. Female subject of child bearing potential who do not agree to remain abstinent or use medically acceptable methods of contraception during the study therapy and for 4 weeks after the end of study therapy.
11. Pregnant / Lactating women.
12. Subject on systemic or oral steroids, oral contraceptive pills or estrogen replacement therapy.
13. Subjects having hypersensitivity to any of the trial drug.
14. Subjects who have completed participation in any other clinical trial during the past six (06) months.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
OBJECTIVE PARAMETERS | Change from Baseline at End of trial [3 month]
  1. Blood sugar fasting in Milligrams per decilitre
OBJECTIVE PARAMETERS | Change from Baseline at End of trial [3 month]
  Blood sugar post prandial Milligrams per decilitre
OBJECTIVE PARAMETERS | Change from Baseline at End of trial [3 month]
  Glycosylated Haemoglobin (HbA1c in %)

SECONDARY OUTCOMES:
SUBJECTIVE PARAMETERS | Change from Baseline at End of trial [3 month]
  Polyurea (excessive urine) grading from 0 to 3
SUBJECTIVE PARAMETERS | Change from Baseline at End of trial [3 month]
  Unclear / turbid urine grading from 0 to 3
SUBJECTIVE PARAMETERS | Change from Baseline at End of trial [3 month]
  Polyphagia( excessive hunger) grading from 0 to 3
SUBJECTIVE PARAMETERS | Change from Baseline at End of trial [3 month]
  Polydipsia (excessive thirst) grading from 0 to 3
SUBJECTIVE PARAMETERS | Change from Baseline at End of trial [3 month]
  Exhaustion / tiredness grading from 0 to 3
SUBJECTIVE PARAMETERS | Change from Baseline at End of trial [3 month]
  Polyneuritis (numbness / tingling/ burning of soles) grading from 0 to 3
SUBJECTIVE PARAMETERS | Change from Baseline at End of trial [3 month]
  Cramps while walking/calf muscle pain grading from 0 to 3
SUBJECTIVE PARAMETERS | Change from Baseline at End of trial [3 month]
  Constipation grading from 0 to 3
SUBJECTIVE PARAMETERS | Change from Baseline at End of trial [3 month]
  Excessive Sweating grading from 0 to 3
SUBJECTIVE PARAMETERS | Change from Baseline at End of trial [3 month]
  Excessive Sleeping grading from 0 to 3
SUBJECTIVE PARAMETERS | Change from Baseline at End of trial [3 month]
  DSQ grading from 0 to 3

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Richa Bhardwaj, M.D. (Ayu.), Principal Investigator — A & U Tibbia College
Locations (1):
- A and U Tibbia College, Delhi, India

IPD SHARING:
Plan to Share IPD: No